CLINICAL TRIAL: NCT05798871
Title: Impact of Erythritol Air-polishing as a Sole Treatment in the Initial Healing of Shallow Periodontal Pockets
Brief Title: Efficacy of Subgingival Erythritol Air Polishing in Treatment of Periodontal Pockets
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Hayder Raad Abdulbaqi, principal investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 746622
Record Dates: First submitted 2023-03-19; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Periodontal Diseases
Keywords: Periodontal Disease; Air-Polishing; Air Abrasion; Periodontitis; Tooth Polishing; periodontal pockets
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Periodontal Pocket

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subgingival erythritol air polishing (Active Comparator): The treatment will include the following therapy steps:
  1. Supragingival debridement.
  2. Subgingival erythritol air polishing by perioflow.
  Interventions: Procedure: Subgingival erythritol air polishing
- Conventional root planing (Active Comparator): The treatment will include the following therapy steps:
  1. Supragingival debridement.
  2. Subgingival root planing by curette.
  Interventions: Procedure: Conventional root planing

INTERVENTIONS:
Procedure: Subgingival erythritol air polishing — The intervention will start with supragingival debridement followed by subgingival erythritol air polishing by perioflow.
  subgingival debridement
  Arms: Subgingival erythritol air polishing
Procedure: Conventional root planing — The intervention will start with supragingival debridement followed by root planing by curette.
  Arms: Conventional root planing

SUMMARY:
Periodontitis is an inflammation associated with destruction of the periodontium that ultimately, if not treated, leads to tooth loss. Clinically, it is characterized by clinical attachment loss (CAL) and bleeding on probing (BOP) accompanied by increased probing pocket depth (PPD) and/or gingival recession. The standard periodontitis treatment aims to restore the homeostasis of the immune system by mechanically reducing the microbial load to levels that are compatible with stability and health. This is achieved by professional mechanical biofilm control and motivation of the patient for oral hygiene measures in order to control the biofilm and avoid disease recurrence. Conventional scaling and root planing (SRP), and air polishing therapy are tools used for professional biofilm control. More recently, air-polishing devices have become a promising alternative to conventional SRP in reducing the clinical time and causing less discomfort and pain for the patients. The objective of this study is to evaluate the efficacy of subgingival erythritol air polishing for initial periodontal pocket healing.

DETAILED DESCRIPTION:
Periodontitis results from a polymicrobial dysbiosis with keystone pathogens affecting the virulence of the entire biofilm community. Thus, the inability of the host immune system to eliminate the biofilm insult leads to a complex chronic response with the destruction of bone and periodontal ligament attachment. The main goal of periodontal therapy is to arrest further attachment loss and, consequently, prevent further disease progression and subsequent tooth loss. In most cases, this goal can be predictably achieved by means of non-surgical periodontal therapy using hand, ultrasonic instruments and air polishing devices. Treatment with scaling and root planing often results in an additional increase of root hypersensitivity, thus impairing the patient's quality of life. Minimally invasive periodontal therapy primarily focus on calculus removal and effective removal of the biofilm rather than on excessive and intentional removal of root cementum.

Air polishing with erythritol powder seems more effective than manual instrumentation at disrupting biofilm in both shallow and deep pockets, whilst it is more gentle on the root surface and soft tissues, and allowing proper attachment of periodontal ligament fibroblasts.

Erythritol powder air-polishing with ultrasonic debridement has reported to need less time than ultrasonic debridement with polishing during periodontal therapy.Therefore, this study will evaluate the impact of erythritol air polishing in resolving periodontal pockets.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be medically healthy with periodontitis.
* Participants should have generalized periodontitis with pockets of PPD = 4 to 6 mm of any stage, unstable, and grade A to C.
* Only teeth with single root will be included.

Exclusion Criteria:

* Participants who have active cavity caries, endodontic treatment.
* Participants who have ongoing orthodontic treatment.
* Participants who have been on antibiotics within the past 4 months.
* Participants who require prophylactic antibiotic coverage.
* Participants who have been on systemic or topical non-steroidal anti- inflammatory drugs for the past 4 months.
* Participants who are pregnant or intended to and lactating mother.
* Participants who have heart valve replacement and have known intolerance or allergy to mouth rinses.
* Participants who have any systemic disease and smokers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-03-05 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Pocket depth | 1 month
  Change of pocket depth (in mm) one month after treatment

SECONDARY OUTCOMES:
Clinical attachment loss | 1 month
  Change of clinical attachment loss (in mm) one month after treatment.
Mean relative changes in beta catenin levels in gingival crevicular fluid. | 1 month
  Mean relative changes in beta catenin levels in gingival crevicular fluid one month after treatment.
Mean relative changes in 8-hydroxy-deoxyguanosine (8-OHdG) levels in gingival crevicular fluid | 1 month
  Mean relative changes in 8-hydroxy-deoxyguanosine (8-OHdG) levels in gingival crevicular fluid one month after treatment
Plaque index | 1 month
  Change in plaque index percentage one month after treatment
Bleeding on probing | 1 month
  Change in bleeding on p[robing percentage one month after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen K Abbass, Principal Investigator — University of Baghdad
Locations (1):
- Hayder R Abdulbaqi, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aljaberi M, Abdulbaqi HR. Efficacy of Erythritol Air Polishing for Inducing Initial Healing of Shallow-to-Moderate Periodontal Pockets and Restoring Gingival Crevicular Fluid beta-Catenin, 8-Hydroxy-Deoxyguanosine and Total Antioxidant Capacity: A Split-Mouth Randomised Clinical Trial. Int J Dent Hyg. 2025 Aug;23(3):559-569. doi: 10.1111/idh.12887. Epub 2024 Dec 17. PMID 39686830